CLINICAL TRIAL: NCT05375071
Title: Use of Blood Flow Restriction (BFR) Therapy in Peri-operative Rehabilitation Following Biceps Tendon Rupture and Medial Patellofemoral Ligament Reconstruction
Brief Title: BFR After Biceps Tendon Repair and MPFLR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Mayo Clinic, study never started
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-006791
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Patellofemoral Joint Dislocation; Bicep Tendon Rupture
Keywords: Bicep tendon repair; medial patellofemoral ligament reconstruction
MeSH Terms: conditions — Patellar Dislocation | interventions — Therapeutics; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation plus blood flow restriction (BFR) therapy (Experimental): Following standard of care surgery, subjects will immediately be started in standard of care physical therapy. Additionally, a BFR Cuff will be applied during physical therapy.
  Interventions: Other: Blood Flow Restriction (BFR) Therapy
- Conventional rehabilitation (Active Comparator): Following standard of care surgery, subjects will immediately be started in standard of care physical therapy.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Blood Flow Restriction (BFR) Therapy — BFR Cuff will be applied to the most proximal portion of the affected arm or leg, immediately before performing exercises during physical therapy. The cuff will remain on for the entire time while an exercise is performed and will be removed in between exercises while the subject rests.
  Arms: Conventional rehabilitation plus blood flow restriction (BFR) therapy
Other: Physical Therapy — Standard of care physical therapy consisting of a structured program progressing from range of motion to strength training and then functional tests
  Arms: Conventional rehabilitation

SUMMARY:
The purpose of this study is to examine the effect of utilizing blood flow restriction (BFR) therapy after distal biceps tendon repair or medial patellofemoral ligament reconstruction (MPFLR) following a tear.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from our ambulatory sports medicine clinics. We will include patients aged 18-80 who suffered a biceps tear and are undergoing biceps repair or MPFLR

Exclusion Criteria:

* Subjects will be excluded if they are undergoing revision biceps repair or revision MPFLR, history of DVT, neurovascular injury, unable to tolerate BFR treatment, unable to complete physical therapy, peripheral vascular disease
* Subjects will be withdrawn from the study if they are unable to tolerate the BFR therapy. Additionally if they suffer from any complications of the therapy they will be withdrawn immediately. This will be facilitated by describing the reasons for withdrawal to the patient prior to initiating the study and ask patients and other providers to inform the investigators if there are any issues or concerns.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Change in strength | Post-operative 6 weeks, 12 weeks, 16 weeks, and 6 months
  Measured by a dynamometer

SECONDARY OUTCOMES:
Change in range of motion | Post-operative 6 weeks, 12 weeks, 16 weeks, and 6 months
  Measured by a goniometer reported in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Kelechi Okoroha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials